CLINICAL TRIAL: NCT02495493
Title: S-1 Plus Cisplatin-based Chemoradiotherapy After Induction Chemotherapy for Locally Advanced Gastric Adenocarcinoma : Phase II Trial
Brief Title: S-1, Cisplatin-based Chemoradiotherapy, Induction Chemotherapy, Locally Advanced Gastric Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sun Young Rha, Severance Hospital, Yonsei University Health System, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0548
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction DCS chemotherapy (Experimental): 1. Induction chemotherapy -- S-1 35mg/m2 bid day 1-14
     * Docetaxel 30 mg/m2 day1, 8
     * Cisplatin 30 mg/m2 day1, 8
  2. Chemoradiotherapy : S-1 20 mg/m2 bid (Day 1-14, 21-28) cisplatin (30 mg/m2/day, Day 1,8, 21,28), Radiotherapy 45 Gy
  Interventions: Drug: Induction DCS chemotherapy

INTERVENTIONS:
Drug: Induction DCS chemotherapy — docetaxel /cisplatin/S-1 followed by chemoradiotherapy (S-1/cisplatin)

SUMMARY:
Currently, for further improved survival outcome, new cytotoxic compounds such as irinotecan and docetaxel have been combined with 5-FU/cisplatin. However, triplet regimen often burdened with higher toxicity and serious neutropenic infection. Therefore, future trials in neoadjuvant and adjuvant settings need to incorporate new molecular agents which improve efficacy, but less toxicity.

DETAILED DESCRIPTION:
Though a significant decrease in its incidence over the last 70 years, gastric cancer remains a significant health problem worldwide. Despite the R0 resection and adjuvant chemotherapy, the prognosis for patients with locally advanced GC remains poor, with 5-year survival rate below 60%. Therefore, active strategy to improve survival outcome is ongoing in gastric cancer. Due to the nature of gastric surgery, postsurgical recovery can be avoided by the administration of systemic therapy and/or radiation prior to the surgical procedure. Furthermore, preoperative therapy has the theoretical advantage of treating an untouched tumor (lack of treatment-induced resistance), with intact vascularization and without fibrotic remodeling of the tumor bed due to surgical trauma. These considerations addressed clinical trials incorporating neoadjuvant treatment for gastric cancer.

Preoperative chemotherapy proved superiority to surgery alone in esophagogastric junction cancer Regarding the pattern of failure, locoregional recurrence after surgical resection has been reported 20-50% of cases. To improve local control and survival outcome, chemoradiotherapy in the neoadjuvant or preoperative setting has been widely applied. In recently published meta-analysis, preoperative chemoradiotherapy combined with surgery significantly reduced the 5-year death rate compared to surgery alone (OR 0.57, P=0.001). Ajani et al reported phase II preoperative chemoradiotherapy (5-fluorouracil/cisplatin and 45 Gy radiotherapy) for localized gastric cancer. Among the 34 stage II/III gastric cancer patients, 30% had pathologic complete response and 24% had pathologic partial response (<10% residual carcinoma). Lowy et al also demonstrated 11% and 63% of complete, partial pathologic responses and preoperative chemoradiotherapy was safe and well tolerated. Based on those rationale, 28 clinical trials with neoadjuvant chemotherapy is ongoing for gastric cancer (clinicaltrial.gov) and the investigators' center is also conducting neoadjuvant chemoradiotherapy trial for localized gastric cancer (NCT01269255).Currently, for further improved survival outcome, new cytotoxic compounds such as irinotecan and docetaxel have been combined with 5-FU/cisplatin. However, triplet regimen often burdened with higher toxicity and serious neutropenic infection. Therefore, future trials in neoadjuvant and adjuvant settings need to incorporate new molecular agents which improve efficacy, but less toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric cancer
* Clinical stage : - Borrmann type IV

  * Large Borrmann type III (>8cm)
  * Locally extensive nodal disease
* No evidence of metastasis
* Patients with tumor lesions which can be easily obtained fresh tumor tissue through repeated biopsies.
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.
* Age≥ 20 years old.
* Performance status of Eastern Cooperative Oncology Group 0 to 2.
* Adequate organ function.

Exclusion Criteria:

1. metastatic disease
2. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
3. Subjects with an uncontrolled major cardiovascular disease (including AMI within 12 months, unstable angina within 6 months, over NYHA class III congestive heart failure, congenital long QT syndrome, 2° or more AV Block and uncontrolled hypertension)
4. Pregnant or lactating female
5. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2019-04 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
pathologic response rate | 12 weeks

SECONDARY OUTCOMES:
overall survival | 3,6,9, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Rha, Principal Investigator — Severance Hosiptal, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Yonsei Cancer Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HS, Koom WS, Baek SE, Kim HI, Jung M, Beom SH, Kang B, Kim H, Chang JS, Choi YY, Son T, Cheong JH, Noh SH, Kim EH, Park JC, Shin SK, Lee SK, Lee YC, Shin SJ, Chung H, Jung I, Chung HC, Lim JS, Hyung WJ, Rha SY. Phase II trial of preoperative sequential chemotherapy followed by chemoradiotherapy for high-risk gastric cancer. Radiother Oncol. 2019 Nov;140:143-149. doi: 10.1016/j.radonc.2019.06.029. Epub 2019 Jul 11. PMID 31302344